CLINICAL TRIAL: NCT01651351
Title: A Phase 4 Double-Blind Study to Assess the Safety and Tolerability of Intravenous Administration of GLASSIA in Healthy Adult Volunteers
Brief Title: GLASSIA Infusion Rate Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 471201
Record Dates: First submitted 2012-07-23; First posted 2012-07-27 (Estimated); Results first posted 2014-05-29 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Alpha1-antitrypsin Deficiency; Healthy Volunteers
Keywords: for this study; volunteers; Focus; Condition:
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Disease | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Day 1:
  * GLASSIA at 0.04 mL/kg/min
  * Placebo at 0.2 mL/kg/min
  Day 15:
  * GLASSIA at 0.2 mL/kg/min
  * Placebo at 0.04 mL/kg/min
  Interventions: Biological: Alpha1-proteinase inhibitor; Biological: Placebo: Human albumin 2.5%
- Cohort 2 (Experimental): Day 1:
  * GLASSIA at 0.2 mL/kg/min
  * Placebo at 0.04 mL/kg/min
  Day 15:
  * GLASSIA at 0.04 mL/kg/min
  * Placebo at 0.2 mL/kg/min
  Interventions: Biological: Alpha1-proteinase inhibitor; Biological: Placebo: Human albumin 2.5%

INTERVENTIONS:
Biological: Alpha1-proteinase inhibitor — GLASSIA will be supplied as a sterile, non-pyrogenic, ready-to-use solution, in single dose 50 mL vials; for intravenous administration.
  Other Names: GLASSIA
Biological: Placebo: Human albumin 2.5% — Intravenous administration

SUMMARY:
The purpose of this study was to generate sufficient safety and tolerability information in support of an increase in the infusion rate of intravenous GLASSIA in the prescribing information from 0.04 to 0.2 mL/kg/min.

DETAILED DESCRIPTION:
To achieve proper masking, 30 participants were randomly assigned to receive either GLASSIA at 0.04 mL/kg/min with a simultaneous administration of placebo (2.5% human albumin in normal saline) at 0.2 mL/kg/min (Cohort 1) or GLASSIA at 0.2 mL/kg/min with a simultaneous administration of placebo at 0.04 mL/kg/min (Cohort 2) on Day 1.

Two weeks later (Day 15), the same participants received the second infusion with the opposite rate of GLASSIA infusion and the corresponding masking placebo infusion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 65 years of age inclusive, at the time of screening
* Body mass index (BMI) in the range of 19.0 to 32.0 kg/m2 (inclusive) and body weight >= 50 kg at the time of screening
* Healthy subject with no clinical evidence of acute and/or chronic disease and no clinically significant abnormalities on hematology panel, clinical chemistry panel, urinalysis, or electrocardiogram (ECG) at the time of screening
* Negative drug screen test at screening. Subject must agree to refrain from heavy alcohol consumption (defined as more than 2 drinks per day on a regular basis) and use of narcotic drugs or illegal substances for at least 2 weeks prior to screening and throughout the course of the study. Subject must also agree to drug screen testing at the discretion of the investigator at any time during the course of the study.
* If female of childbearing potential, subject presents with a negative serum pregnancy test and agrees to employ adequate birth control measures for the duration of the study
* If male, the subject must agree to use an acceptable form of birth control throughout the study and for at least 90 days after dosing. Additionally, the subject must agree to abstain from sperm donation for 90 days after the last administration of investigational product.
* Subject is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Known history of OR positive serological evidence at the time of screening for hepatitis A virus (HAV), hepatitis B virus (HBV), hepatitis C virus (HCV), Parvovirus B19 (PVB19) or human immunodeficiency virus (HIV) type 1/2 infection
* Known history of hypersensitivity or adverse reactions (e.g. urticaria, breathing difficulty, severe hypotension, or anaphylaxis) following administration of blood or blood components
* Documented immunoglobulin A (IgA) deficiency (<7 mg/dL at screening)
* Evidence of uncontrolled hypertension (systolic blood pressure of >160 mm Hg, and/or diastolic blood pressure of >100 mm Hg despite anti-hypertensive medications)
* Subject is nursing or intends to begin nursing during the course of the study
* Subject has participated in a clinical trial and has received an investigational product within 60 days prior to screening
* Subject has a planned medical procedure within the study period
* Any clinically significant medical, psychiatric, or cognitive illness or recreational drug/alcohol use that, in the opinion of the investigator, may impede the subject's ability to comply with the study procedures, pose increased risk to the subject's safety, or confound the interpretation of study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07-31 (Actual); Primary Completion 2013-01-16 (Actual); Study Completion 2013-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Overland Park, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted in the U.S at 1 study site. The first participant was enrolled in July 2012.
Pre-assignment Details: Thirty five healthy potential participants were enrolled at the clinical study site. Four were screen failures, and one was a back up participant who did not participate. Therefore, 30 participants were randomized.
Groups:
- Cohort 1: Day 1: - GLASSIA at 0.04 mL/kg/min - Placebo at 0.2 mL/kg/min Day 15: - GLASSIA at 0.2 mL/kg/min - Placebo at 0.04 mL/kg/min Alpha1-proteinase inhibitor: GLASSIA will be supplied as a sterile, non-pyrogenic, ready-to-use solution, in single dose 50 mL vials; for intravenous administration. Placebo: Human albumin 2.5%: Intravenous administration
- Cohort 2: Day 1: - GLASSIA at 0.2 mL/kg/min - Placebo at 0.04 mL/kg/min Day 15: - GLASSIA at 0.04 mL/kg/min - Placebo at 0.2 mL/kg/min Alpha1-proteinase inhibitor: GLASSIA will be supplied as a sterile, non-pyrogenic, ready-to-use solution, in single dose 50 mL vials; for intravenous administration. Placebo: Human albumin 2.5%: Intravenous administration
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Cohort 1: Day 1: - GLASSIA at 0.04 mL/kg/min - Placebo at 0.2 mL/kg/min Day 15: - GLASSIA at 0.2 mL/kg/min - Placebo at 0.04 mL/kg/min Placebo: Human albumin 2.5%: Intravenous administration
- Cohort 2: Day 1: - GLASSIA at 0.2 mL/kg/min - Placebo at 0.04 mL/kg/min Day 15: - GLASSIA at 0.04 mL/kg/min - Placebo at 0.2 mL/kg/min Placebo: Human albumin 2.5%: Intravenous administration
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (8) | 29 (13) | 28 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 12 | 11 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Infusions Associated With a Reduction in Infusion Rate or Discontinuation of Infusion Due to an Adverse Event (Regardless of Adverse Event Causality Assessment)
Time Frame: Day 1 and Day 15
Population: Safety Analysis Set
Measure: Number; unit: Infusions
Arm/Group | GLASSIA at 0.04 mL/kg/Min + Placebo at 0.2 mL/kg/Min | GLASSIA at 0.2 mL/kg/Min + Placebo at 0.04 mL/kg/Min
Number analyzed (Participants) | 30 | 30
Infusions | 0 | 0

2. Secondary Outcome: Number of Infusions With Temporally Associated Adverse Events (AEs) That Began During or Within 1 Hour of Infusion Completion
Description: Number of infusions with temporally associated AEs with an onset time during or within 1 hour of infusion completion, regardless of causality assessment
Time Frame: Within 1 hour of infusion completion
Population: Safety Analysis Set
Measure: Number; unit: Infusions
Arm/Group | GLASSIA at 0.04 mL/kg/Min + Placebo at 0.2 mL/kg/Min | GLASSIA at 0.2 mL/kg/Min + Placebo at 0.04 mL/kg/Min
Number analyzed (Participants) | 30 | 30
Infusions | 3 | 1

3. Secondary Outcome: Number of Infusions With Temporally Associated Adverse Events (AEs) That Began During or Within 24 Hours of Completion of an Infusion
Description: Number of infusions with temporally associated AEs with an onset time during or within 24 hours of infusion completion, regardless of causality assessment
Time Frame: Within 24 hours of the end of infusion
Population: Safety Analysis Set
Measure: Number; unit: Infusions
Arm/Group | GLASSIA at 0.04 mL/kg/Min + Placebo at 0.2 mL/kg/Min | GLASSIA at 0.2 mL/kg/Min + Placebo at 0.04 mL/kg/Min
Number analyzed (Participants) | 30 | 30
Infusions | 5 | 3

4. Secondary Outcome: Number of Infusions With Temporally Associated Adverse Events (AEs) That Began During or Within 72 Hours of Completion of an Infusion
Description: Number of infusions with temporally associated AEs with an onset time during or within 72 hours of infusion completion, regardless of causality assessment
Time Frame: Within 72 hours of the end of infusion
Population: Safety Analysis Set
Measure: Number; unit: Infusions
Arm/Group | GLASSIA at 0.04 mL/kg/Min + Placebo at 0.2 mL/kg/Min | GLASSIA at 0.2 mL/kg/Min + Placebo at 0.04 mL/kg/Min
Number analyzed (Participants) | 30 | 30
Infusions | 7 | 5

5. Secondary Outcome: Number of Possibly or Probably Related Adverse Events (AEs) That Began During an Infusion
Description: Number of AEs that occurred during an infusion and were deemed related to study product administration
Time Frame: Day 1 and Day 15
Population: Safety Analysis Set
Measure: Number; unit: adverse events
Arm/Group | GLASSIA at 0.04 mL/kg/Min + Placebo at 0.2 mL/kg/Min | GLASSIA at 0.2 mL/kg/Min + Placebo at 0.04 mL/kg/Min
Number analyzed (Participants) | 30 | 30
adverse events | 1 | 0

6. Secondary Outcome: Number of Possibly or Probably Related Adverse Events That Occurred Between 72 Hours and 14 Days After Infusion
Description: Number of AEs that occurred between 72 hours and 14 day following an infusion and were deemed related to study product administration
Time Frame: 72 hours post infusion to 14 days post infusion
Population: Safety Analysis Set
Measure: Number; unit: adverse events
Arm/Group | GLASSIA at 0.04 mL/kg/Min + Placebo at 0.2 mL/kg/Min | GLASSIA at 0.2 mL/kg/Min + Placebo at 0.04 mL/kg/Min
Number analyzed (Participants) | 30 | 30
adverse events | 0 | 0

7. Secondary Outcome: Number of Participants Testing Positive for Hepatitis A Virus (HAV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Parvovirus B19 (PVB19) or Human Immunodeficiency Virus (HIV) Following Treatment With GLASSIA
Description: Number of participants with seroconversion
Time Frame: 105 days
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
participants
  HAV | 0
  HBV | 0
  HCV | 0
  PVB19 | 0
  HIV | 0

ADVERSE EVENTS:
Time Frame: Throughout the study period of 105 days per participant
Groups:
- GLASSIA Infusion Rate- 0.04 mL/kg/Min: Participants who received simultaneous infusions of: - GLASSIA at 0.04 mL/kg/min - Placebo at 0.2 mL/kg/min
- GLASSIA Infusion Rate- 0.2 mL/kg/Min: Participants who received simultaneous infusions of: - GLASSIA at 0.2 mL/kg/min - Placebo at 0.04 mL/kg/min
Arm/Group | GLASSIA Infusion Rate- 0.04 mL/kg/Min | GLASSIA Infusion Rate- 0.2 mL/kg/Min
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 8/30 | 4/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLASSIA Infusion Rate- 0.04 mL/kg/Min (N=30) | GLASSIA Infusion Rate- 0.2 mL/kg/Min (N=30)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 6 (7) | 3 (5)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
Simultaneous infusion of GLASSIA and placebo did not allow adverse events (AEs) to be unquestionably ascribed to either one. Any observed AE which was assessed by the investigator as related to treatment was conservatively attributed to GLASSIA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may not publish without the prior written consent of Sponsor